CLINICAL TRIAL: NCT06981676
Title: The Developmental Origins of Obesity: Effect of Maternal Supplementation With Polyunsaturated Fatty Acids and Insights Into Adipose and Immune Progenitor Cells
Brief Title: The Developmental Origins of Obesity
Acronym: OMEGA-Stem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Paola Casanello Toledo, Full Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1221812
Record Dates: First submitted 2025-01-20; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Maternal Obesity; Obesity
Keywords: Pregestational Obesity; Maternal Obesity; Omega 3; PUFAs; LCPUFAs
MeSH Terms: conditions — Pregnancy in Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Normalweight Group (NW) (No Intervention): Pregnant women with normal weight and pregnancy usual care
- NW plus PUFAs group (Experimental): NW women, supplemented with high levels of PUFA (600 mg/day DHA/EPA).
  Interventions: Dietary Supplement: DHA and EPA
- Pregestational obesity Group (PGO) (No Intervention): Pregnant women with PGO and pregnancy usual care
- Pregestational obesity Group (PGO) plus PUFAs group (Experimental): Women with PGO with high PUFA supplementation (600 mg/day DHA/EPA)
  Interventions: Dietary Supplement: DHA and EPA

INTERVENTIONS:
Dietary Supplement: DHA and EPA — Women will receive daily supplementation of LCPUFAs (DHA and EPA) from first trimester until delivery
  Arms: NW plus PUFAs group; Pregestational obesity Group (PGO) plus PUFAs group

SUMMARY:
Pregestational obesity (PGO, BMI ≥30) is a significant independent risk factor for the development of obesity in childhood and adolescence. Notably, elevated levels of IL-6 and leptin have been found in the cord blood of offspring born to women with PGO, along with increased body fat. Both our research and that of others have shown an upregulation of pro-inflammatory genes in cord blood monocytes and alterations in innate immune function, including a blunted response to pro-inflammatory stimuli. However, it remains unclear whether these effects are due to an altered immune response in differentiated immune cells or if they are programmed earlier in gestation, during the progenitor cell stage.

Long-chain polyunsaturated fatty acids (LCPUFAs) are crucial for cellular function, acting as precursors to membrane components and signaling molecules involved in cardiovascular, metabolic, and immune processes. Modern dietary patterns have led to a relative deficiency in n-3 LCPUFAs, such as Docosahexaenoic acid (DHA) and Eicosapentaenoic acid (EPA). As a result, international health guidelines recommend LCPUFA supplementation during pregnancy. Studies have shown that increased intake of n-3 LCPUFAs during pregnancy exerts effective anti-inflammatory effects in the maternal circulation, adipose tissue, and placenta.

The recently completed MIGHT study (NCT02574767), which involved 1005 women with overweight or PGO, investigated the effects of DHA supplementation during pregnancy (200 mg vs. 800 mg/day). A subgroup of the newborns from this cohort also participated in the EpiFat study (NCT04249635), conducted by our team (2017-2021). The findings demonstrated that maternal DHA supplementation (800 mg/day) significantly reduced body fat and improved adipose metabolic markers in offspring at birth, with these effects persisting until 4 months of age. Additionally, the cord blood monocytes of PGO offspring exhibited increased expression of pro-inflammatory genes (IL-6, MCP-1, TNF-α, IL-8), but these effects were completely reversed in the offspring of DHA-supplemented women. These results provide strong evidence of pro-inflammatory programming in innate immune cells and adiposity in offspring of women with PGO, and show that maternal PUFA supplementation during pregnancy can reverse these early obesity biomarkers. However, it remains unclear whether these effects persist into early childhood (5 years of age), particularly in high-risk populations such as those born to women with PGO.

Moreover, we hypothesize that maternal obesogenic signals during early embryonic development may affect the progenitor cells of adipocytes (mesenchymal stem cells, MSC) and monocytes (hematopoietic stem cells, HSC), potentially leading to long-term effects on the offspring.

This study hypothesizes that: "Maternal obesity increases the risk of childhood obesity by programming adipose and immune progenitor cells, an effect that may be mitigated by maternal supplementation with polyunsaturated fatty acids during pregnancy." To test this hypothesis, we propose:

A pilot clinical study to examine whether maternal PGO affects the lineage commitment, number, TLR4 signaling, and epigenetic markers (ChIP-seq) of monocyte (HSC) and adipocyte (MSC) progenitor cells, and whether maternal supplementation with PUFAs during pregnancy can modify these effects. The OMEGA Stem study will invite 160 healthy women (80 with normal weight and 80 with pregestational obesity) with singleton pregnancies to participate. Participants will receive either 600 mg/day of EPA/DHA (1 capsule) or standard antenatal care. A trained midwife will enroll the women <16 weeks of pregnancy, with data collection (sociodemographic information, clinical data and blood samples) at study initiation, 26-28 weeks, and at delivery. Neonatal body composition will be assessed by a trained midwife (24-48 hours after delivery) through anthropometric measurements and skinfold thickness, calculated using Catalano's formula.

DETAILED DESCRIPTION:
Epidemiological evidence recognizes pregestational obesity (PGO) as an independent risk factor in the development of maternal complications and adverse perinatal outcomes, including preeclampsia, gestational diabetes, neonatal intensive care unit admission, among others. A recent study using data from 162,129 mothers and their children from 37 maternal-infant cohorts concluded that 21.7- 41.7% of childhood overweight/obesity prevalence could be attributed to maternal overweight and obesity together. The link between early exposures during development and an increased risk of developing chronic diseases in later life was named "Fetal programming" by Professor David Barker, and is currently called Developmental Origins of Health and Disease (DOHaD). Today there is clear evidence in humans and animals that not only in utero under-nutrition but also over-nutrition increases the cardiometabolic risk in the offspring. However, new efforts are required to clarify the mechanisms by which maternal obesity before and during pregnancy impinges on an increased risk of chronic disease in the progeny.

This project has the following General aim Evaluate if the supplementation with PUFAs during pregnancy in women with obesity affects the molecular markers of lineage commitment in adipose (MSC) and immune (HSC) progenitor cells of their offspring and if these correlate with adiposity and inflammatory immune markers at birth.

2.1- To determine if PGO modifies the number of HSC in cord blood at birth and their lineage commitment (myeloid vs lymphoid) and the effect of maternal supplementation with PUFAs during pregnancy.

2.2- To evaluate if there is an altered expression and activation of the LPS/TLR4/AKT pathway in cord blood HSPCs from women with PGO and if maternal PUFA supplementation modifies these responses.

2.3- To determine if PGO and DHA supplementation affect the PPARγ-dependent adipogenic commitment in WJ-derived MSC from their offspring at birth.

2.4- To evaluate if maternal PGO confers the signature of trained epigenetic markers (histones and DNA methylation profile) in HSC/MSC and if maternal DHA supplementation changes these epigenetic memory hallmarks.

2.5- To determine if maternal PGO and supplementation with PUFAs during pregnancy affects the early adiposity markers (body composition, and metabolic markers) and immune phenotype (monocytes and T cells) in their offspring at birth.

METHODOLOGY This pilot study (maternal Obesity steM cEll programming; OMEGA Stem) is conceived to interrogate the progenitor cells of both monocytes (HSPC) and adipocytes (MSC) of the offspring of women with PGO who received PUFA supplements during pregnancy. For this purpose, 160 women (80 normal weight and 80 PGO) are invited to participate in a pilot study of n-3 PUFA supplementation in pregnancy and stem cell markers in their offspring. Once they consent, they will be given capsules of EPA/DHA 600 mg/day or the standard antenatal care.

The participants are women who seek prenatal care in the Red de Salud UC-Christus, in Santiago Chile. The inclusion criteria are: first prenatal visit <14 weeks gestation, pregestational BMI between 18.5 and 24.9 for the NW groups, and BMI >30 for the PGO groups, have singleton pregnancy, ≥18 years of age and plan to deliver at the Hospital Clínico UC- Christus or San Carlos de Apoquindo Clinic in Santiago de Chile. The exclusion criteria are: preexisting diabetes, GDM, preeclampsia, multiple gestations, chronic cardio-respiratory disorder or neurological o genetic defects of the fetus, history of an eating disorder, food allergy, any high-risk pregnancy condition (MINSAL 2015).

Participant recruitment will proceed as follows:

The obstetrician will introduce the project to women who meet the inclusion criteria and provide them with an informative flyer. A midwife will then follow up with a phone call to explain the project's details and offer an invitation to participate. Additional information will be available on a dedicated website, where any interested woman can submit a form to request more details and provide contact information. For those who meet the inclusion criteria, a midwife will reach out to invite them to join the project.

After the informed consent process, the women who agree to participate are enrolled. Enrolled women will be randomized to receive supplementation of LCPUFAs or the standard prenatal care. Four groups, of 40 women each, will be formed according to their pregestational BMI (at < 14 weeks of gestation) and the n-3 PUFAs supplementation

1. Normal weight Group (NW): NW women who receive standard prenatal care.
2. NW+PUFA Group: NW women who receive supplements with high levels of PUFA (600 mg/day DHA/EPA).
3. Pregestational obesity Group (PGO): women with PGO who receive standard prenatal care.
4. PGO+PUFA Group: women with PGO who receive supplements with high levels of PUFA.

Outcomes The primary outcome of this pilot study is the effect of DHA on maternal obesity-induced adipogenic and myelopoietic commitment and epigenetic and metabolic programming of the neonatal progenitor cells (HSC & MSC).

The secondary outcomes are:

The effect of DHA on PGO-induced a) changes in the number of HSC in cord blood, b) changes in LPS/TLR/AKT pathway activation in HSC, and c) the presence of epigenetic hallmarks of trained immunity in these stem cells at birth.

Variables Newborn and maternal variables of the study will be homologous to those analyzed for the MIGHT and EPIFAT studies.

Clinical evaluations and follow up: a trained Midwife will follow up the patients by phone and coordinate the follow up visit at 26-28 weeks of gestation.

In the first and follow up visit, midwife collect clinical data, measure height and weight, take blood samples and apply the Chilean Mediterranean Diet Survey.

At the delivery, the clinical team in the hospital collect maternal blood, cord blood samples and the placenta.

24- 48 hours after delivery a trained Midwife visits the woman and the newborn, collects the delivery clinical data and performs the neonatal body composition assessment through anthropometrics and skinfold determinations.

Compliance with the supplementation: maternal blood samples are collected at baseline, at 26-28 weeks of gestation and at the delivery. Plasma and red blood cell PUFA levels will be evaluated to assess compliance. Moreover at the 3rd-trimester visit (26-28 weeks) and in the delivery participants will be asked to bring the empty bottles and remaining capsules which will be counted and registered to calculate adherence.

Dropouts: participants who consume <50% of the n-3 PUFA capsules or participants allocated to the reference group who report > 300 mg n-3 LC-PUFA intake will be considered dropouts. The intervention will be discontinued in women who present obstetric or medical complications.

Sample size: for the metabolic programming of the neonatal stem cells (principal outcome), we have considered the mean difference of 0.90 in this variable described by González et al., power of 80% and p-value of 0.05. The estimation of sample size (STATA software) is 25 subjects per group and considering a 20% of loss to follow up, and an extra 20% of loss at delivery, the adjusted sample size is 32 subjects per group.

Ethics: The study will be performed in accordance with the Helsinki Declaration, and written informed consent will be obtained from all participants during pregnancy (Institutional Ethics Committee submission #210624014).

In vitro studies:

Umbilical cord blood and umbilical cord will be collected at delivery in Terumo collecting bags (50-100 ml) and stored at room T° until processing. The umbilical cord, will be stored at 4°C. Both samples will be transported to the lab (200 mt distance from maternity ward) in the next 30-45 minutes after delivery. Whole Cord blood and HSC isolation & characterization. Whole blood (2 ml) will be used to stimulate & immunophenotype monocytes by FACS as classical, non-classical, and intermediate subsets and T cell immunophenotyped (Th1, Th2, Th17, Treg). Cord Blood Mononuclear Cells (CBMCs) will be obtained by ficoll gradient, as described27. HSCs CD34+ will be isolated from 200×106 freshly isolated CBMCs using positive immunomagnetic sorting with microbeads (Miltenyi). HSCs will be analyzed by FACS for purity as CD34+CD38- and HPCs as CD34+CD38lo and lineage commitment markers evaluated. Wharton´s Jelly-derived MSC will be isolated as previously described108. Briefly, the umbilical cord will be cut in slices, and 2 mm2 pieces of WJ will be obtained and set as explants in 6 well plates and cultured in DMEM with 10 % FBS and antibiotics. WJ-MSC will be immunophenotyped by flow cytometry to evaluate the presence of surface proteins of MSC lineage as CD73, CD44, CD90, CD29 and CD105, and the absence of hematopoietic markers CD45, CD34, CD14 and lack of HLA-D(see collaboration letter Prof Harmsen in Annexes). Adipogenesis will be induced for up to 4 days in an adipogenic induction cocktail medium (low-glucose DMEM, 5% FBS, 1 mM dexamethasone, 200 mmol/L indomethacin, 500 mmol/L 3-isobutyl-1-methylxanthine, 170 pmol/L insulin, and 0.13 penicillin/streptomycin) and adipogenic phenotype analyzed through PPARγ expression64. Quantification of proteins, cytokines, metabolic markers in maternal/neonatal plasma. Glycemia, insulin, lipid profile, Leptin, Adiponectin and hepatic enzymes will be measured in the clinical lab at PUC. Inflammatory cytokines and mediators (TNF-α, IL-6, IL-1β, MCP-1, IL-10) will be determined by Cytometric Beads Array (CBA) Flex Set (BD Bioscience) as published. Proteins (TLR4, PI3K, AKT, pAKT, PPARγ) in HSC and MSC will be measured by flow cytometry. qPCR for gene expression. RNA will be isolated from HSC, MSC, and monocytes using a commercial kit (RNeasy Qiagen). RT will be performed (ImProm-II-RT System, Promega). QPCR will be carried out using oligonucleotide primers for target genes (TNFα, IL-6, Il-1β, MCP-1, and IL-10). GADPH, ATP5F1, and RPLP2 will be used as internal references. Relative expression of target genes will be calculated with the method of 2-delta CT, as published. Chromatin Immunoprecipitation-sequencing. Whole-genome ChIP-seq for H3K27ac, H3K4me3, and H3K4me1 in primary HSC & MSC will be performed using iDeal ChIP-seq kit for Histones (Diagenode). DNA methylation analysis. DNA methylation status in peripheral monocytes in the infants will be analyzed using the EPIC 850k (Illumina) as used with EpiFat at birth. Data analysis was performed using a Bioconductor packaged workflow (version 3.13) to analyze methylation matrices. Fatty acid profile analysis. Quantitative extraction/separation of total lipids from maternal at two moments during pregnancy (before and 14-20 weeks after supplementation), and cord blood plasma and RBCs will be performed according to the method of Bligh & Dyer, and published. Analysis of FA methyl-esters (FAME) will be performed in plasma and RBC samples as published. Sample size will be by convenience (and preliminary results), and for the primary outcomes in HSCs and MSCs a n=30 per group was estimated. Statistical analysis. For descriptive statistics mean ± SD or median and IQ range for quantitative variables, and % with n for categories will be used. Distributions will be verified with a Shapiro Wilk test, ANOVA or Kruskal Wallis to evaluate differences between groups and Spearman/Pearson correlation to determine the association between dependent/independent variables. Independent variables will be fitted to logistic/lineal regression models to evaluate interactions or identify confounding factors. For in vitro studies, comparisons between two or more groups will be performed by Student's t-test and ANOVA, respectively, and post hoc Dunns or Bonferroni. STATA/Graphpad Prism will be used, considering p<0.05 as a cut-off for significance.

ELIGIBILITY:
Inclusion Criteria:

* First prenatal visit <14 weeks gestation
* Pregestational BMI between 18.5 and 24.9 for the NW groups and BMI >30 for the PGO groups,
* To have singleton pregnancy,
* ≥18 years of age and plan to deliver at the Hospital Clínico UC- Christus

Exclusion Criteria:

* Preexisting diabetes
* GDM
* Preeclampsia,
* Multiple gestations
* Chronic cardio-respiratory disorder or neurological o genetic defects of the fetus
* History of an eating disorder, food allergy,
* Any high-risk pregnancy condition (MINSAL 2015)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
PPARγ gene expression in mesenchymal stem cells isolated from the umbilical cord of newborns from normal-weight and obese mothers supplemented or not with DHA | At birth
  Adipogenic commitment will be assessed by qPCR measuring the expression of PPARγ. Unit of measure: PPARg gene expression (RQ-fold change) in mesenchymal cells
Myelopoietic commitment of hematopoietic stem cells (HSC) from umbilical cord blood of newborns from normal-weight and obese mothers supplemented or not with DHA | At birth
  Myelopoietic commitment will be assessed by flow cytometry, identifying the expression of CD38 in CD34+ HSC. Unit of Measure: Percentage (%) and Mean fluorescence intensity (MFI) of CD38 in HSC (CD34+ cells)

SECONDARY OUTCOMES:
Number of CD34+ hematopoietic stem cells (HSC) in cord blood. | At birth
  The number of CD34+ HSC will be quantified by flow cytometry. Unit of Measure: Number of CD34+ cells per mL of cord blood.
Activation of LPS/TLR4/AKT pathway in hematopoietic stem cells (HSC). | At birth
  Activation of this pathway will be assessed by measuring phosphorylated AKT (pAKT) levels by flow cytometry in CD34+ HSC. Unit of Measure: Mean fluorescence intensity (MFI)
Presence of "trained immunity epigenetic hallmarks" in hematopoietic stem cells (HSC). | At birth
  The presence of specific histone modifications (H3K27ac, H3K4me3, H3K4me1) will be assessed by Chromatin Immunoprecipitation-sequencing in CD34+ HSC. Unit of Measure: Name of genes (DNAseq) that present these epigenetic marks.

OTHER OUTCOMES:
Neonatal fat mass at birth | 24 - 48 hours after birth
  Neonatal fat mass (grams) will be calculated through anthropometric measurements (weight, length), and flank skinfold (calibrated Harpenden caliper) using Catalano's formula.
  Unit of Measure: Fat mass (grams) = 0.39055 (weight) + 0.0453 (Flank skinfold) - 0.03237 (Length) + 0.54657, as published by Catalano et al., Am J Obstetrics Gynecology 1995.

CONTACTS AND LOCATIONS:
Locations (1):
- Red Salud UC Christus Hospital, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided